CLINICAL TRIAL: NCT03331341
Title: A Pilot Trial of Adriamycin, Pembrolizumab, Vinblastine, and Dacarbazine (APVD) for Patients With Untreated Classical Hodgkin Lymphoma
Brief Title: Doxorubicin Hydrochloride, Pembrolizumab, Vinblastine, and Dacarbazine in Treating Patients With Classical Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Ryan Lynch, Associate Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9805; NCI-2017-01718 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9805 (Other: Fred Hutch/University of Washington Cancer Consortium); RG1001581 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Classical Hodgkin Lymphoma
Keywords: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Dacarbazine; Doxorubicin; pembrolizumab; Vinblastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (APVD) (Experimental): PART A: Patients receive doxorubicin hydrochloride intravenously (IV), vinblastine IV, and dacarbazine IV on days 1 and 15. Patients also receive pembrolizumab IV over 30 minutes on days 1 and 22 of cycle 1 and on day 15 of cycle 2. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  PART B: Patients receive doxorubicin hydrochloride IV, vinblastine IV, dacarbazine IV, and pembrolizumab IV as in part A, but undergo a total of 6 treatment cycles.
  Interventions: Drug: Dacarbazine; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Drug: Vinblastine

INTERVENTIONS:
Drug: Dacarbazine — Given IV
  Other Names: 4-(Dimethyltriazeno)imidazole-5-carboxamide; 5-(Dimethyltriazeno)imidazole-4-carboxamide; Asercit; Biocarbazine; Dacarbazina; Dacarbazina Almirall; Dacarbazine - DTIC; Dacatic; Dakarbazin; Deticene; Detimedac; DIC; Dimethyl (triazeno) imidazolecarboxamide; Dimethyl Triazeno Imidazol Carboxamide; Dimethyl Triazeno Imidazole Carboxamide; dimethyl-triazeno-imidazole carboxamide; Dimethyl-triazeno-imidazole-carboximide; DTIC; DTIC-Dome; Fauldetic; Imidazole Carboxamide; Imidazole Carboxamide Dimethyltriazeno; WR-139007
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Drug: Vinblastine — Given IV
  Other Names: Vincaleucoblastine; VLB

SUMMARY:
This phase II trial studies the side effects of doxorubicin hydrochloride, pembrolizumab, vinblastine, and dacarbazine in treating patients with classical Hodgkin lymphoma. Drugs used in chemotherapy, such as doxorubicin hydrochloride, vinblastine, and dacarbazine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with pembrolizumab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Giving doxorubicin hydrochloride, pembrolizumab, vinblastine, and dacarbazine may work better in treating classical Hodgkin lymphoma.

DETAILED DESCRIPTION:
OUTLINE:

PART A: Patients receive doxorubicin hydrochloride intravenously (IV), vinblastine IV, and dacarbazine IV on days 1 and 15. Patients also receive pembrolizumab IV over 30 minutes on days 1 and 22 of cycle 1 and on day 15 of cycle 2. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.

PART B: Patients receive doxorubicin hydrochloride IV, vinblastine IV, dacarbazine IV, and pembrolizumab IV as in part A, but undergo a total of 6 treatment cycles.

After completion of study treatment, patients are followed up at 30 days and then up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have cHL that has not been previously treated

  * Part A: Any stage
  * Part B: Must be stage 3 or 4
* Patients must be appropriate candidates for at least 2 cycles of doxorubicin hydrochloride (adriamycin), bleomycin, vinblastine and dacarbazine (ABVD) (6 cycles for Part B patients) or doxorubicin hydrochloride, vinblastine, dacarbazine (AVD) (this could include patients ranging from favorable risk early stage disease to poor prognosis advanced stage disease)
* Patients must have measurable FDG-avid disease defined by standard criteria (Lugano 2014) and a minimum of 1.0 cm in diameter
* Patients should not have evidence of active central nervous system lymphoma
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients must have a left ventricular ejection (LVEF) >= 50% within 56 days of enrollment
* Patients must have adequate labs within 10 days of treatment
* Absolute neutrophil count (ANC) >= 1,500/mm^3 (without transfusion or growth factor support)
* Platelets >= 100,000/mm^3 (without transfusion or growth factor support)
* Hemoglobin >= 8 g/dL. Growth factor and/or transfusion support is permissible to stabilize participant prior to study treatment if needed. There is no lower limit to cytopenias if related to bone marrow involvement
* Serum creatinine < 1.5 mg/dl or creatinine clearance greater than 30/ml per minute by Cockcroft Gault formula
* Total bilirubin =< 1.5 times upper limit of normal OR direct bilirubin =< upper limit of normal (ULN) for participants with total bilirubin levels > 1.5 x ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 times upper limit of normal (=< 5 x ULN for participants with liver metastases)
* All patients must be informed of the investigational nature of this study and have given written consent in accordance with institutional and federal guidelines
* Patients must be anticipated to complete all planned study therapy
* Male subjects should agree to use an adequate method of barrier contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year

Exclusion Criteria:

* Patients known positive for human immunodeficiency virus (HIV), or infectious hepatitis type B or C
* Pregnant or nursing women; men or women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Patients with other prior malignancies except for adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, breast or cervical cancer in situ, or other cancer from which the patient has been disease-free for 5 years or greater, unless approved by the protocol chair or co-chair
* Patients who have other medical conditions that would contraindicate treatment with aggressive chemotherapy (including active infection, uncontrolled hypertension, congestive heart failure, unstable angina pectoris, or myocardial infarction within the past 6 months, uncontrolled arrhythmia, severe pulmonary disease or requirement of supplemental oxygen)
* Active ischemic heart disease or congestive heart failure
* Concurrent use of other anti-cancer agents or experimental treatments
* Known current or prior autoimmune disease with the exception of vitiligo
* Active or prior history of pneumonitis/interstitial lung disease that required corticosteroids
* Current use of supplemental oxygen
* Is known to have received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of trial treatment. Administration of killed vaccines is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Lynch, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lynch RC, Ujjani CS, Poh C, Warren EH, Smith SD, Shadman M, Till B, Raghunathan VM, Alig S, Alizadeh AA, Gulhane A, Chen DL, Tseng Y, Coye H, Shelby M, Ottemiller S, Keo S, Verni K, Du H, Vandermeer J, Gaston A, Rasmussen H, Martin P, Marzbani E, Voutsinas J, Gopal AK. Concurrent pembrolizumab with AVD for untreated classic Hodgkin lymphoma. Blood. 2023 May 25;141(21):2576-2586. doi: 10.1182/blood.2022019254. PMID 36913694

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (APVD): PART A: Patients receive doxorubicin hydrochloride intravenously (IV), vinblastine IV, and dacarbazine IV on days 1 and 15. Patients also receive pembrolizumab IV over 30 minutes on days 1 and 22 of cycle 1 and on day 15 of cycle 2. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity.
  PART B: Patients receive doxorubicin hydrochloride IV, vinblastine IV, dacarbazine IV, and pembrolizumab IV as in part A, but undergo a total of 6 treatment cycles.
  Dacarbazine: Given IV
  Doxorubicin Hydrochloride: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given IV
  Vinblastine: Given IV
Period: Overall Study
Arm/Group | Treatment (APVD)
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (APVD)
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 40
  More than one race | 1
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: PART A: Number of Participants Who Complete of 2 Cycles of Adriamycin, Pembrolizumab, Vinblastine and Dacarbazine (APVD)
Description: Number of participants who complete 2 cycles of treatment without a dose delay of >3 weeks. Toxicity leading to dose delay will be assessed using CTCAE v5.0.
Time Frame: At the end of Cycle 2 (each cycle is 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (APVD)
Number analyzed (Participants) | 30
Participants | 30

2. Primary Outcome: PART B: Event Free Survival at 1 Year
Description: Number of participants who are event free at 1 year. An event is defined as progression, biopsy proven recurrence, initiation of next line of chemotherapy, or death.
Time Frame: At the end of 1 year after completing 2 cycles of treatment (each cycle is 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (APVD)
Number analyzed (Participants) | 50
Participants | 49

3. Secondary Outcome: Proportion of Fludeoxyglucose F-18 (FDG)-Positron Emission Tomography PET2 Negative (Deauville Score 1-3) Patients After 2 Cycles of APVD
Description: The Deauville 5 point scale is scored as follows: 1, no uptake above background; 2, uptake ≤ mediastinum; 3, uptake > mediastinum but ≤ liver; 4, uptake moderately > liver; 5, uptake markedly higher than liver and/or new lesions; X, new areas of uptake unlikely to be related to lymphoma.
Time Frame: After 2 cycles (each cycle is 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (APVD)
Number analyzed (Participants) | 49
Participants | 30

ADVERSE EVENTS:
Time Frame: Adverse events are collected beginning with the first dose of treatment through 30 days after last dose, approximately 7 months. All-Cause Mortality was monitored/assessed up to 1 year after completing the 2nd cycle.
Arm/Group | Treatment (APVD)
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 8/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (APVD) (N=50)
Febrile Neutropenia (Blood and lymphatic system disorders) | 5 (8)
Septic Shock (Infections and infestations) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Guillain-Barré syndrome (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (APVD) (N=50)
Abdominal Pain (Gastrointestinal disorders) | 7 (9)
Alanine Aminotransferase Increased (Investigations) | 19 (55)
Alkaline Phosphatase Increased (Investigations) | 5 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (14)
Anemia (Blood and lymphatic system disorders) | 24 (45)
Anxiety (Psychiatric disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8)
Asparate Aminotransferase Increased (Investigations) | 13 (28)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Bloating (Gastrointestinal disorders) | 3 (3)
Blurred Vision (Eye disorders) | 3 (3)
Bone Pain (Musculoskeletal and connective tissue disorders) | 8 (11)
Chills (General disorders) | 8 (8)
Constipation (Gastrointestinal disorders) | 34 (39)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Creatinine increased (Investigations) | 3 (3)
Decreased lymphocytes (Investigations) | 5 (27)
Decreased neutrophil count (Investigations) | 34 (188)
Decreased white blood cells (Investigations) | 5 (21)
Diarrhea (Gastrointestinal disorders) | 14 (17)
Dizziness (Nervous system disorders) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Dysguesia (Nervous system disorders) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Edema (General disorders) | 3 (4)
Fatigue (General disorders) | 24 (27)
Fever (General disorders) | 8 (11)
Flushing (Vascular disorders) | 4 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Headache (Nervous system disorders) | 16 (19)
Hemorrhoids (Gastrointestinal disorders) | 3 (3)
Hot flashes (Vascular disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (6)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (10)
Hypokalemia (Metabolism and nutrition disorders) | 12 (15)
Hyponatremia (Investigations) | 4 (13)
Hypothyroidism (Endocrine disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 13 (13)
Mucositis oral (Gastrointestinal disorders) | 7 (9)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 36 (43)
Neuropathy (Nervous system disorders) | 14 (15)
Night sweats (General disorders) | 3 (3)
Oral pain (Gastrointestinal disorders) | 7 (9)
Pain (General disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5)
Paresthesia (Nervous system disorders) | 7 (7)
Pruritis (Skin and subcutaneous tissue disorders) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 10 (12)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Syncope (Nervous system disorders) | 4 (5)
Upper respiratory infection (Infections and infestations) | 10 (14)
Vomiting (Gastrointestinal disorders) | 14 (22)
White blood count decreased (Investigations) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT03331341/Prot_SAP_000.pdf